CLINICAL TRIAL: NCT01379664
Title: Volatile Anesthetic Choice and Duration of Hospitalization: A Quality Improvement and Cost-control Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Professor & Chair, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-440
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Duration of Hospitalization
Keywords: Sevoflurane; Isoflurane; volatile anesthetic; duration of hospitalization
MeSH Terms: interventions — Isoflurane; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isoflurane (Experimental): Isoflurane is to be administered to patients in this arm during surgery
  Interventions: Drug: Isoflurane
- Sevoflurane (Experimental): Sevoflurane is to be administered to patients in this arm during surgery
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Isoflurane — Isoflurane is administered to patient during surgery as it would normally be administered by the attending anesthesiologist
  Arms: Isoflurane
Drug: Sevoflurane — Sevoflurane is administered to patient during surgery as it would normally be administered by the attending anesthesiologist
  Arms: Sevoflurane

SUMMARY:
Preliminary retrospective data suggest that the relatively soluble but inexpensive volatile anesthesia isoflurane prolongs the duration of hospitalization compared to the less soluble but more expensive anesthetic sevoflurane. Even a small reduction in the duration of hospitalization would easily compensate for the modest additional cost of sevoflurane. The investigators therefore propose to test the primary hypothesis that duration of hospitalization is longer with isoflurane than sevoflurane.

The investigators will also test the secondary hypotheses that: 1) pain scores are greater in patients recovering from isoflurane than sevoflurane anesthesia; and, 2) opioid consumption is greater after isoflurane than sevoflurane anesthesia. All statistical analyses will be adjusted for age, gender, race, baseline risk, 9 and procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must have surgery in G operating room suite

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1584 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isoflurane | Sevoflurane
Started | 714 | 870
Completed | 714 | 870
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isoflurane | Sevoflurane | Total
Number analyzed (Participants) | 714 | 870 | 1584
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (16.5) | 53.6 (16.6) | 53.5 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 408 | 502 | 910
  Male | 306 | 368 | 674

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Isoflurane | Sevoflurane
Number analyzed (Participants) | 714 | 870
Days | 4.9 [2.0 to 8.4] | 4.4 [1.5 to 7.8]
Statistical Analysis 1: Comparison: Isoflurane vs Sevoflurane; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney); Ratio of Geometric Means = 1.06, 95% CI 2-sided [0.97 to 1.16]

2. Secondary Outcome: Time-weighted Average Verbal Rating Pain Score
Description: Time-weighted average VRS (Verbal Rating Scale) pain score over the first 72 h after surgery as recorded by nurses at approximately 4-h intervals. The VRS pain score is from 0 (no pain) to 10 (worst imaginable pain).
Time Frame: up to 72 hours after surgery
Population: Postoperative pain measurements were not available for 19 isoflurane patients and 20 sevoflurane patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Isoflurane | Sevoflurane
Number analyzed (Participants) | 682 | 850
units on a scale | 3.6 (1.9) | 3.6 (1.8)
Statistical Analysis 1: Comparison: Isoflurane vs Sevoflurane; Test type: Superiority or Other; p = 0.87, Generalized estimating equation model; Generalized estimating equation model weighted by inverse propensity score; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.23 to 0.19]

3. Secondary Outcome: Total Intraoperative Opioid Consumption
Description: Total amount of opioid in IV morphine equivalents used during surgeyr
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Isoflurane | Sevoflurane
Number analyzed (Participants) | 714 | 870
mg | 32 (1.3) | 33 (1.6)
Statistical Analysis 1: Comparison: Isoflurane vs Sevoflurane; Test type: Superiority or Other; p = 0.74, Generalized estimating equation model; Generalized estimating equation model weighted by propensity score; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-4.7 to 3.3]

ADVERSE EVENTS:
Arm/Group | Isoflurane | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 0/701 | 0/870
Other Adverse Events (participants affected / at risk) | 0/701 | 0/870

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes